CLINICAL TRIAL: NCT03763240
Title: Effect of BSE on Blood Glucose
Brief Title: BSE on Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BSE
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Blood Glucose, High

STUDY DESIGN:
Intervention Model Description: Parallel arm study with placebo and intervention substance
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each participant receives the kit that corresponds to his/her study ID. The randomization is blind to both participants and the Investigator during the study.
  The randomization list is kept with the local pharmacy during the entire study. Sealed envelopes with randomization information for each participant are send to investigator and may be opened in case of emergency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BSE (Active Comparator): Sulforaphane-containing broccoli sprout extract (BSE). The study product is BSE with standardized amounts of sulforaphane. BSE contains a mixture of maltodextrin as a bulking agent and copper chlorophyllin (E 141) as a food additive. BSE is a dried powder of an aqueous extract of broccoli sprouts that provides a consistent and stable source of sulforaphane.
  Interventions: Dietary Supplement: BSE
- Placebo (Placebo Comparator): A mixture of maltodextrin and copper chlorophyllin will be used as placebo. The active compound and the placebo are the same except BSE. The placebo will look similar to the BSE-containing mixture.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: BSE — BSE powder will be provided as dry mixtures in sealed, non-transparent portion size bags. Each BSE bag contains 150 μmole, equal to 0.26 g, sulforaphane at a minimum. The mixtures are suspended with appr. 1 dl water and are ingested once daily in the morning. BSE should be stored at room temperature in dry conditions.
  The doses of sulforaphane contained in the BSE is not possible to get by eating fresh broccoli, thus it has to be given as an extract.
  Arms: BSE
Dietary Supplement: Placebo — Placebo powder will be provided as dry mixtures in sealed, non-transparent portion size bags. The mixtures are suspended with appr. 1 dl water and are ingested once daily in the morning.
  Arms: Placebo

SUMMARY:
Here we will investigate the effect of sulforaphane, provided as a broccoli sprout extract (BSE) on blood glucose in pre-diabetic individuals without metformin treatment. This will address whether BSE could be used to improve glucose control in drug-naïve pre-diabetic individuals. The participants will receive BSE or placebo in a randomized double-blind parallel arm study. The participants will take their study compound once daily over 12 weeks. The primary study variable is fasting glucose.

DETAILED DESCRIPTION:
Here we will investigate the effect of sulforaphane, provided as a broccoli sprout extract (BSE) on blood glucose in pre-diabetic individuals without metformin treatment. This will address whether BSE could be used to improve glucose control in drug-naïve pre-diabetic individuals. The participants will receive BSE or placebo in a randomized double-blind parallel arm study. The participants will take their study compound once daily over 12 weeks. The primary study variable is fasting glucose.

ELIGIBILITY:
Inclusion Criteria:

* Impaired fasting glucose, defined as fasting blood glucose 6.1-6.9 mM.
* Written informed consent
* Age 35-75 years. Participating women of fertile age must have no current pregnancy, which will be assessed by pregnancy test.
* Body mass index 27-45 kg/m2

Exclusion Criteria:

* Diagnosed with diabetes mellitus according to the WHO criteria
* Anti-diabetic medication
* Active liver disease
* At screening or at any subsequent visit a level of aspartate aminotransferase (ASAT) or alanine aminotransferase (ALAT) of more than three times the upper limit of the normal range
* Gastrointestinal ailments which may interfere with the ability to adequately absorb sulforaphane
* At screening visit creatinine > 130 µmol/L
* Coagulation disorder or current anti-coagulant therapy, which may be affected by the BSE
* Diagnosed with a cardiovascular disease or known cardiovascular event, transient ischemic attack, coronary by-pass surgery or other coronary vessel intervention within 6 months prior to enrolment
* Systemic glucocorticoid treatment
* Herbal treatment, defined as food supplement (except multivitamin treatment) with herbal or vegetable extracts that may affect blood glucose
* Allergy to broccoli
* Participant unable to understand the study information
* Participation in other clinical trial which may affect the outcome of the present study
* Any other physical or psychiatric condition or treatment that in the judgment of the investigator makes it difficult to participate in the study.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
The primary effect variable is venous fasting blood glucose. | 12 weeks
  Participants will be analysed using intraindividual one-tailed comparisons before and after treatment and compared between the placebo and BSE arms

SECONDARY OUTCOMES:
Change of long-term blood glucose concentration measured as glycated hemoglobin at 12 weeks | 12 weeks
  Intraindividual change of long-term blood glucose concentration measured as glycated hemoglobin (HbA1c) in mmol/mol at 12 weeks relative to baseline compared between participants treated with BSE and placebo, respectively.
Change of insulin resistance measured as HOMA-IR at 12 weeks | 12 weeks
  Intraindividual change of insulin resistance measured as Homeostasis model assessment-2 estimates of insulin resistance (HOMA-IR) at 12 weeks relative to baseline compared between participants treated with BSE and placebo, respectively.
Change of insulin secretion measured as HOMA-B at 12 weeks | 12 weeks
  Intraindividual change of insulin secretion measured as Homeostasis model assessment-2 estimates of beta-cell function (HOMA-B) at 12 weeks relative to baseline compared between participants treated with BSE and placebo, respectively.
Change of body mass index at 12 weeks | 12 weeks
  Intraindividual change of body mass index (BMI), measured as the body weight in kilogram divided by the square of the length in meter, at 12 weeks relative to baseline compared between participants treated with BSE and placebo, respectively.
Change of total cholesterol at 12 weeks | 12 weeks
  Intraindividual change of total cholesterol concentration in plasma (measured in mmol/l) at 12 weeks relative to baseline compared between participants treated with BSE and placebo, respectively.
Change of LDL cholesterol at 12 weeks | 12 weeks
  Intraindividual change of low-density lipoprotein (LDL) cholesterol concentration in plasma (measured in mmol/l) at 12 weeks relative to baseline compared between participants treated with BSE and placebo, respectively.
Change of HDL cholesterol at 12 weeks | 12 weeks
  Intraindividual change of high-density lipoprotein (HDL) cholesterol concentration in plasma (measured in mmol/l) at 12 weeks relative to baseline compared between participants treated with BSE and placebo, respectively.
Change of triglycerides at 12 weeks | 12 weeks
  Intraindividual change of serurm triglyceride concentration (measured in mmol/l) at 12 weeks relative to baseline compared between participants treated with BSE and placebo, respectively.
Change of fatty liver index at 12 weeks | 12 weeks
  Intraindividual change of fatty liver index (based on body mass index in kg per square meter, waist circumference in centimeter, triglycerides in mmol/l and gamma-glutamyl transferase in microkat/l) at 12 weeks relative to baseline compared between participants treated with BSE and placebo, respectively.
Change of insulin clearance at 12 weeks | 12 weeks
  Intraindividual change of insulin clearance (measured as fasting plasma C-peptide concentration in nmol/l divided by fasting plasma insulin concentration mIE/l) at 12 weeks relative to baseline compared between participants treated with BSE and placebo, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Gothia Forum, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dwibedi C, Axelsson AS, Abrahamsson B, Fahey JW, Asplund O, Hansson O, Ahlqvist E, Tremaroli V, Backhed F, Rosengren AH. Effect of broccoli sprout extract and baseline gut microbiota on fasting blood glucose in prediabetes: a randomized, placebo-controlled trial. Nat Microbiol. 2025 Mar;10(3):681-693. doi: 10.1038/s41564-025-01932-w. Epub 2025 Feb 10. PMID 39929977